CLINICAL TRIAL: NCT00024245
Title: Phase I and Clinical Pharamcologic Study of 10-Propargyl-10-Deazaaminopterin (PDX) in Combination With Probenecid in Adults With Advanced Solid Tumors
Brief Title: 10-Propargyl-10-Deazaaminopterin Plus Probenecid in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: MSKCC-01014; CDR0000068905 (Registry Identifier: PDQ (Physician Data Query)); NCI-H01-0077
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2003-03

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — 10-propargyl-10-deazaaminopterin; Probenecid

INTERVENTIONS:
Drug: pralatrexate
Drug: probenecid

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Probenecid may increase the effectiveness of 10-propargyl-10-deazaaminopterin by making tumor cells more sensitive to the drug.

PURPOSE: Phase I trial to study the effectiveness of combining 10-propargyl-10-deazaaminopterin and probenecid in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of 10-propargyl-10-deazaaminopterin and probenecid in patients with advanced solid tumors.
* Determine the therapeutic activity of this regimen in these patients.
* Determine the toxic effects of this regimen in these patients.
* Determine the pharmacokinetics of this regimen in these patients.

OUTLINE: This is a dose-escalation study of 10-propargyl-10-deazaaminopterin (PDX) and probenecid.

Patients receive probenecid IV and PDX IV on day 1. Treatment repeats every 2 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive sequentially escalating doses of probenecid and PDX until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 35-40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed cancer that is potentially incurable by standard chemotherapy, radiotherapy, or surgical procedures

  * Failed prior first-line therapy (patients are also eligible if no effective first-line therapy exists)
* Previously treated or clinically stable brain metastases are allowed
* No leukemia or lymphoma
* No clinically significant pleural effusions or ascites

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 4,000/mm^3
* Platelet count at least 160,000/mm^3
* Hemoglobin greater than 10 g/dL
* Serum and RBC folate normal

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* SGOT or SGPT less than 2 times upper limit of normal

Renal:

* Creatinine no greater than 1.2 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No unstable angina
* No congestive heart failure
* No cardiac arrhythmia

Other:

* Homocysteine normal
* No grade III or IV edema
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 6 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy (4 weeks for nitrosoureas or mitomycin) and recovered

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy to bone marrow-containing areas and recovered

Surgery:

* See Disease Characteristics
* No prior pneumonectomy

Other:

* No concurrent folic acid or potentially nephrotoxic agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-05; Study Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naiyer Rizvi, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States